CLINICAL TRIAL: NCT03646136
Title: Benefits of Retained Cystoscopy Fluid Following Benign Laparoscopic and Robotic Hysterectomy; A Randomized Controlled Trial
Brief Title: Post Hysterectomy Benefits of Retained Cystoscopy Fluid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Rachael Bailey Smith, Dr. Rachael Smith, Principal Investigator, University of Arizona
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: UA IRB# 1808885089
Record Dates: First submitted 2018-08-07; First posted 2018-08-24 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Urinary Retention
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: PACU nurses and patients will not be aware of which arm patient was randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retained Cystoscopy Fluid (Experimental): Retained 200mL normal saline used for distending media following completion of diagnostic cystoscopy
  Interventions: Procedure: Retained fluid
- Cystoscopy Fluid Emptied (Active Comparator): Emptied 200mL normal saline used for distending media following completion of diagnostic cystoscopy
  Interventions: Procedure: Emptied fluid

INTERVENTIONS:
Procedure: Retained fluid — Retained fluid
  Arms: Retained Cystoscopy Fluid
Procedure: Emptied fluid — Emptied fluid
  Arms: Cystoscopy Fluid Emptied

SUMMARY:
The purpose of this research study is to compare outcomes for women in two study arms that include retaining the cystoscopy distending fluid after minimally invasive hysterectomy verses completely emptying the cystoscopy distending fluid. The outcomes being measured for research purposes include the time spent to first spontaneous urination after surgery, rate of indwelling catheter insertion, length of recovery room stay, the amount of bladder discomfort immediately postoperative and over the first 24 hours postoperative, bladder symptoms over the first 24 hours postoperative, and patient satisfaction.

DETAILED DESCRIPTION:
Acute urinary retention can be a common postoperative complication following hysterectomy. One of the many benefits of minimally invasive surgery is shorter hospital stay following a major procedure such as laparoscopic or robotic hysterectomy. An important postoperative milestone before discharge from the postoperative anesthesia care unit (PACU) is spontaneous voiding. If unable to spontaneously void due to urinary retention, insertion of an indwelling catheter may be required. Awaiting a spontaneous void in the recovery room can lead to longer hospital and PACU stays, greater cost, and patient dissatisfaction. At the conclusion of traditional laparoscopic or robotic-assisted hysterectomy, intraoperative cystoscopy is performed to evaluate for urologic injury. One possible strategy to more quickly facilitate a postoperative spontaneous void is to retain the cystoscopy distending fluid at conclusion of cystoscopy rather than emptying the bladder of the distending fluid. Although there is no published research investigating voiding time following laparoscopic or robotic hysterectomy using strategies such as backfilling the bladder before removal of the indwelling catheter or retaining the cystoscopy distending fluid following diagnostic cystoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, greater than or equal to 18 years old
* English-speaking
* Undergoing laparoscopic or robotic hysterectomy for benign indications by one of the three minimally invasive gynecologic surgeons at Banner University Medical Center - Phoenix.

Exclusion Criteria:

* Preoperative indications of pelvic organ prolapse
* Preoperative indications of urinary incontinence
* Lower urologic (bladder or ureteric) injury identified at time of hysterectomy or during intraoperative cystoscopy
* Patients given any measure to aid in visualization of ureteral patency including dextrose, phenazopyridine, indigo carmine, methylene blue, sodium fluorescein, or furosemide.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women undergoing minimally invasive hysterectomy.
Enrollment: 120 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Time to spontaneous void | From surgery end time up to 4 hours
  Measure of time to spontaneous urination in the recovery room post hysterectomy. Time of urination is measured by the recovery room nurse from surgery end time.

SECONDARY OUTCOMES:
Foley catheter insertion rate | 2 weeks
  Rate of patient's requiring Foley catheter insertion post hysterectomy if unable to spontaneously void in recovery room or anytime within 2 weeks postoperative.
Length of recovery room stay | From time of randomization up to 12 hours postoperative
  Measure of time from surgery end time to discharge home from the recovery room post hysterectomy.
4-Item Patient Satisfaction Measure | 12 hours
  Self reported patient satisfaction survey related to ability to urinate in the recovery room, amount of time given to urinate, amount of time it took to urinate, and overall bladder discomfort. Each item is scored 1-5 (1=very satisfied, 5=very dissatisfied).
2-Item Patient Satisfaction Measure | 24 hours
  Self reported patient satisfaction survey related to voiding function over 24 hours and overall bladder discomfort over 24 hours. Each item is scored 1-5 (1=very satisfied, 5=very dissatisfied).
3-Item Bladder Symptoms Measure | 24 hours
  Self reported bladder symptom measure of burning, frequency, and urgency with voiding over the 24 hours postoperative. Measured as Yes/No.
2-Item Bladder pain Measure | 12 hours
  Self reported bladder pain intensity on initial arrival to the recovery room and at discharge from the recovery room. Each item is scored 1-10 (1=no discomfort, 10=most discomfort).
3-Item Bladder pain Measure | 24 hours
  Self reported bladder pain intensity over 24 hours postoperative, bladder discomfort before urination, and bladder discomfort after urination. Each item is scored 1-10 (1=no discomfort, 10=most discomfort).

CONTACTS AND LOCATIONS:
Overall Officials: Rachael Smith, DO, Principal Investigator — UofA College of Medicine Dept of OBG/Banner University Medical Center Phoenix
Locations (1):
- Banner University Medical Center Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ellahi A, Stewart F, Kidd EA, Griffiths R, Fernandez R, Omar MI. Strategies for the removal of short-term indwelling urethral catheters in adults. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD004011. doi: 10.1002/14651858.CD004011.pub4. PMID 34184246
- [Derived] Smith RB, Mahnert ND, Hu C, Steck-Bayat K, Womack AS, Mourad J. Impact of Retained Cystoscopy Fluid after Laparoscopic Hysterectomy: A Randomized Controlled Trial. J Minim Invasive Gynecol. 2021 Feb;28(2):288-296. doi: 10.1016/j.jmig.2020.05.024. Epub 2020 Jun 4. PMID 32505857